CLINICAL TRIAL: NCT02329392
Title: Assessment of Skin Perfusion Pressure as an Indicator of Tissue Oxygenation in Cardiac Surgery Patients Undergoing Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2014-0070
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral Circulation During On-pump Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SPP: Patients undergoing cardiac surgery with perioperative monitoring of Skin Perfusion Pressure

SUMMARY:
This study is aim to evaluate usefulness of the perioperative monitoring of skin perfusion pressure as an indicator of perpheral perfusion in patients undergoing on-pump cardiac surgery. Association of the intraoperative and postoperative 6hr skin perfusion pressure with perioperative serum lactate level is going to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 yrs, scheduled for elective on-pump cardiac surgery

Exclusion Criteria:

* known peripheral arterial occlusive disease, patients without swan ganz catheter insertion, heart transplantation, infective endocarditis, emergency surgery, hemodynamic instability requiring vasopressor, preoperative lactate > 2mmol/L, known liver cirrhosis, pregnant, cognitive dysfunction, being unable to communicate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patinets > 20 years old who are scheduled for elective on-pump cardiac surgery
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment of skin perfusion pressure | From post induction to 6 hours

SECONDARY OUTCOMES:
Assessment of arterial lactate level | From post induction to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea